CLINICAL TRIAL: NCT02491866
Title: Development and Implementation of a Computerized Adaptative Testing (CAT) of Self-perceived Quality of Care in Psychiatry
Brief Title: Computerized Adaptative Testing of Self-perceived Quality of Care in Psychiatry
Acronym: QDSPsyCAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-22
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- psychiatric patients (Other): patients with schizophrenia, bipolar disorder or depression according DSM V criteria
  Interventions: Other: to develop and validate a Computerized Adaptative Testing

INTERVENTIONS:
Other: to develop and validate a Computerized Adaptative Testing — * Elaboration of a pool of items, based on literature review and interview with patients.
  * Selection of the most relevant items based on a qualitative approach using cognitive interview with patients.
  * Calibration of the item bank : the psychometric properties of the item bank will be based on classical test and item response theories and approaches, including the evaluation of unidimensionality, item response theory model fitting, and analyses of differential item functioning.
  * Metrological validation of the CAT.
  * Analysis of the implementation of the CAT in clinical practice using interview with professionals and patients.

SUMMARY:
Objectives

1. to develop and validate a Computerized Adaptative Testing (CAT) of self-perceived quality of care in Psychiatry.
2. to analyze the implementation of this new measure in clinical practice : qualitative analysis of the relationship patient/professional.

DETAILED DESCRIPTION:
Prospective and multicentric study

1. Development and validation of the CAT. 4 steps :

   * Elaboration of a pool of items, based on literature review and interview with patients.
   * Selection of the most relevant items based on a qualitative approach using cognitive interview with patients.
   * Calibration of the item bank : the psychometric properties of the item bank will be based on classical test and item response theories and approaches, including the evaluation of unidimensionality, item response theory model fitting, and analyses of differential item functioning.
   * Metrological validation of the CAT.
2. Analysis of the implementation of the CAT in clinical practice using interview with professionals and patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia, bipolar disorder or depression according DSM V
* criteria
* age over 18 years
* informed consent to participate
* French as the native language

Exclusion Criteria:

* diagnosis other than schizophrenia, bipolar disorder or depression according DSM V criteria
* decompensated organic disease, and mental retardation

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1400 (Estimated)
Dates: Start 2015-05-27 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Quality of care | 19 months
  computerized Adaptative Testing

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hopital de la conception Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Fernandes S, Brousse Y, Zendjidjian X, Cano D, Riedberger J, Llorca PM, Samalin L, Dassa D, Trichard C, Laprevote V, Sauvaget A, Abbar M, Misdrahi D, Berna F, Lancon C, Coulon N, El-Hage W, Rozier PE, Benoit M, Giordana B, Caqueo-Urizar A, Yon DK, Tran B, Auquier P, Fond G, Boyer L. Psychometric Assessment of an Item Bank for Adaptive Testing on Patient-Reported Experience of Care Environment for Severe Mental Illness: Validation Study. JMIR Ment Health. 2024 May 16;11:e49916. doi: 10.2196/49916. PMID 38753416
- [Derived] Boyer L, Fernandes S, Brousse Y, Zendjidjian X, Cano D, Riedberger J, Llorca PM, Samalin L, Dassa D, Trichard C, Laprevote V, Sauvaget A, Abbar M, Misdrahi D, Berna F, Lancon C, Coulon N, El-Hage W, Rozier PE, Benoit M, Giordana B, Caqueo-Urizar A, Yon DK, Tran B, Auquier P, Fond G. Development of the PREMIUM computerized adaptive testing for measuring the access and care coordination for patients with severe mental illness. Psychiatry Res. 2023 Oct;328:115444. doi: 10.1016/j.psychres.2023.115444. Epub 2023 Sep 1. PMID 37677894
- [Derived] Fernandes S, Fond G, Zendjidjian X, Michel P, Lancon C, Berna F, Schurhoff F, Aouizerate B, Henry C, Etain B, Samalin L, Leboyer M, Misdrahi D, Llorca PM, Coldefy M, Auquier P, Baumstarck K, Boyer L. A conceptual framework to develop a patient-reported experience measure of the quality of mental health care: a qualitative study of the PREMIUM project in France. J Mark Access Health Policy. 2021 Feb 23;9(1):1885789. doi: 10.1080/20016689.2021.1885789. PMID 33680364
- [Derived] Fernandes S, Fond G, Zendjidjian XY, Baumstarck K, Lancon C, Berna F, Schurhoff F, Aouizerate B, Henry C, Etain B, Samalin L, Leboyer M, Llorca PM, Coldefy M, Auquier P, Boyer L; French PREMIUM Group. Measuring the Patient Experience of Mental Health Care: A Systematic and Critical Review of Patient-Reported Experience Measures. Patient Prefer Adherence. 2020 Nov 3;14:2147-2161. doi: 10.2147/PPA.S255264. eCollection 2020. PMID 33192054
- [Derived] Fernandes S, Fond G, Zendjidjian X, Michel P, Baumstarck K, Lancon C, Berna F, Schurhoff F, Aouizerate B, Henry C, Etain B, Samalin L, Leboyer M, Llorca PM, Coldefy M, Auquier P, Boyer L. The Patient-Reported Experience Measure for Improving qUality of care in Mental health (PREMIUM) project in France: study protocol for the development and implementation strategy. Patient Prefer Adherence. 2019 Jan 21;13:165-177. doi: 10.2147/PPA.S172100. eCollection 2019. PMID 30718945